CLINICAL TRIAL: NCT01302145
Title: A Double-blind, Randomized, Placebo-controlled, Parallel Design Study, in Patients With Type 2 Diabetes Mellitus, to Investigate the Safety, Pharmacokinetics and Pharmacodynamics Interactions of Multiple Oral Doses of ASP1941 and Metformin
Brief Title: Drug to Drug Interaction Study With ASP1941 and Metformin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1941-CL-0056; 2007-005614-39 (EudraCT Number)
Record Dates: First submitted 2011-02-21; First posted 2011-02-23 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: pharmacokinetics; metformin; Drug to drug interaction; ASP1941
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ipragliflozin; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASP1941 + metformin (Experimental): Oral
  Interventions: Drug: ASP1941; Drug: Metformin
- Placebo + metformin (Placebo Comparator): Oral
  Interventions: Drug: Metformin; Drug: Placebo

INTERVENTIONS:
Drug: ASP1941 — Tablet
  Arms: ASP1941 + metformin
Drug: Metformin — Tablet
Drug: Placebo — Tablet
  Arms: Placebo + metformin

SUMMARY:
A study to investigate the effect on safety, pharmacokinetics and pharmacodynamics when ASP1941 is administered as add-on therapy to metformin.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes
* Stable disease under metformin monotherapy (between 1500-3000

mg/day) or dual therapy with metformin (1500-3000 mg/day) and a Sulfonylureum Derivative (SUD) for at least 3 months

* Fasting Serum Glucose: 7-11.5 mmol/l (after wash-out)
* Stable Fasting Blood Glucose (FBG) at the end of wash-out
* BMI between 18.5 and 40.0 kg/m2, inclusive

Exclusion Criteria:

* Subjects with type 1 diabetes
* Any diabetes related macro-complications, painful diabetic neuropathy, diabetic macular edema or diabetic proliferative retinopathy
* Clinical significant renal disease (CLcr <60 ml/min as assessed during a 24h creatinine clearance on Day-2
* Recent evidence (e.g. within the last 6 months) of severe hypoglycemia, for example plasma glucose <3 mmol/l (<55 mg/dl) or requiring hospitalization
* Pulse <40 or >90; Systolic Blood Pressure >160 mmHg; Diastolic Blood Pressure > 100 mmHg

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-02-25 (Actual); Primary Completion 2009-12-09 (Actual); Study Completion 2009-12-09 (Actual)

PRIMARY OUTCOMES:
Safety assessed by incidence of adverse events, vital signs, 12-lead ECG and glucose monitoring | 5 weeks

SECONDARY OUTCOMES:
Pharmacodynamics assessed by serum glucose change | 5 weeks
Pharmacokinetics assessed by metformin plasma concentration change | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Europe B.V.
Locations (5):
- Hungary (2):
  - Balatonfüred
  - Budapest
- Groningen, Netherlands
- Warsaw, Poland
- Bratislava, Slovakia

REFERENCES:
- [Derived] Veltkamp SA, van Dijk J, Collins C, van Bruijnsvoort M, Kadokura T, Smulders RA. Combination treatment with ipragliflozin and metformin: a randomized, double-blind, placebo-controlled study in patients with type 2 diabetes mellitus. Clin Ther. 2012 Aug;34(8):1761-71. doi: 10.1016/j.clinthera.2012.06.027. Epub 2012 Jul 15. PMID 22795925
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=5